CLINICAL TRIAL: NCT02537080
Title: The Effect of Nimodipine in the Preoperative Period on the Onset of Postoperative Cognitive Dysfunction in Adults
Brief Title: The Effect of Nimodipine on the Postoperative Cognitive Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: higher POCD in nimodipine Group
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, Vlasta Dostalova, MD, PhD, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201508-S22P
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Postoperative cognitive dysfunction; Nimodipin; Anesthesia
MeSH Terms: conditions — Cognitive Dysfunction; Postoperative Cognitive Complications | interventions — Nimodipine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nimodipine group (Experimental): 1 tbl of 30 mg nimodipine will be administered orally with premedication
  Interventions: Drug: Nimodipine group
- Control group (Experimental): 1 tbl of placebo will be administered orally with premedication
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Nimodipine group — the stability of the blood pressure will be managed in interval plus minus 15% of patient's resting blood pressure
  Other Names: nimodipine
  Arms: Nimodipine group
Drug: Control group — the stability of the blood pressure will be managed in interval plus minus 15% of patient's resting blood pressure
  Other Names: placebo
  Arms: Control group

SUMMARY:
The calcium channel blocker nimodipine dilates cerebral blood vessels and can pass through the blood-brain barrier, providing neuroprotective effects by selectively improving cerebral blood flow and inhibiting neuronal necrosis and apoptosis. Nimodipine significantly inhibited the production of tumor necrosis factor TNF-α and interleukin IL-1β, and also of nitric oxide and prostaglandin E2 from lipopolysaccharide-stimulated microglia. Abnormal cytokine networks are important in the development of nerve cell damage that leads to cognitive impairment.

DETAILED DESCRIPTION:
All patients aged above 60 years undergoing planned neurosurgical operations in the duration up to 4 hours under general anesthesia will be included in the study. The patients will not be sedated by any type of benzodiazepine. A dose of 30 mg nimodipine or placebo will be applied 45 minutes before the surgery according to the randomization. Anesthesia will be managed according to the standardised protocol. Concentration of desflurane will be adjusted according to entropy values (target 40-50). Analgetics will be applied according to surgical pleth index (SPI) values. Sufentanil will not be applied in the last 15 minutes. Extubation will be performed at the operating theatre when meeting all extubation criteria including train of four ratio (TOFR) above 92%. Neither syntophylline, nor pharmacological decurarization (syntostigmine) will be applied to the patients.During the surgery, blood pressure will be maintained within ± 15% of the patient's normal blood pressure. Cognitive dysfunction tests will be executed on the day before the surgery, two hours after the surgery and on the third postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* Glascow coma scale GCS 15 preoperatively
* American Society of Anesthesiologists ASA risk I - III
* planned brain surgery
* duration of procedure up to 4 hours.

Exclusion Criteria:

* blood pressure below 130/80 torr preoperatively
* previous vascular surgery
* concomitant use of antiepileptic drugs, rifampicin
* allergy to nimodipine
* known liver cirrhosis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in cognitive behavior | within the first 3 days after surgery
  measured by Addenbrooks cognitive test

CONTACTS AND LOCATIONS:
Overall Officials: Vlasta Dostalova, MD, PhD, Study Director — University Hospital Hradec Kralove
Locations (1):
- University Hospital, Hradec Králové, Czechia